CLINICAL TRIAL: NCT06758102
Title: Assessing the Impact of a 12-week Dance Intervention on Quality of Life, Post-surgical Pain, Fatigue, and Body Image in Breast Cancer Survivors
Brief Title: Dance Study for Post-surgical Pain in Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-586
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Survivorship; Pain, Postoperative
Keywords: Breast Cancer Survivorship; Breast Cancer Survivor; Survivorship; Pain, Postoperative; PPSP; Persistent Post-Surgical Pain
MeSH Terms: conditions — Breast Neoplasms; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dance Program (Experimental): 30 enrolled participants will complete the following:
  * Baseline in-person or virtual visit with surveys.
  * 12 weekly virtual dance classes.
  * Follow up in-person or virtual visit with post-intervention surveys.
  Interventions: Behavioral: Dance Program

INTERVENTIONS:
Behavioral: Dance Program — A 12-week, virtual dance program consisting of seated and standing choreography and contemporary style elements will be taught by a certified dance instructor. Sessions will be conducted by the HIPAA-compliant, video-conferencing platform, Zoom.

SUMMARY:
The purpose of this study is to examine how a 12-week, virtual dance program may improve pain and quality of life in participants with persistent post-surgical pain, or PPSP, following mastectomy or lumpectomy.

DETAILED DESCRIPTION:
This is a single-arm, Phase 1 study is to assess how a 12-week, virtual dance program may improve persistent post-surgical pain (PPSP) and other participant-reported outcomes of quality of life, fatigue, and body image for breast cancer survivors following mastectomy or lumpectomy.

The study procedures including screening for eligibility and surveys.

Participation in this research study is expected to last up to 16 weeks.

It is expected that about 30 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* History of Stage 0-III invasive breast cancer
* Having undergone lumpectomy or mastectomy
* Moderate to severe persistent post-surgical pain, as defined by pain scores ≥3 on a numerical rating scale (NRS) of 0-10 (10 being the most severe pain) at least 3 months after completion of surgery, chemotherapy, and/or radiation
* Pain scores of 3-4 are categorized as moderate pain; scores of 5-10 are categorized as severe pain26
* Age ≥ 18 years
* Able to read and understand English (to complete required questionnaires and participate in classes)
* Ability to provide informed consent
* Ability to perform seated exercises

Exclusion Criteria:

* Unstable cardiovascular disease in the last 6 months
* Psychiatric disorders or conditions that would preclude participation in the study intervention (e.g. untreated major depression or psychosis, untreated substance use disorder, severe personality disorder)
* Metastatic breast or other concurrent cancer
* Pregnant
* Recent history of attending regular dance or similar classes (e.g. yoga or tai chi classes i.e. 20 or more classes in the past 6 months)
* Planned surgery anticipated during the intervention period
* History of a chronic medical condition that has the potential to significantly impact upper extremity function (e.g. stroke, Parkinson's disease, Multiple Sclerosis)
* Currently enrolled in a physical therapy course
* Presence of medical conditions or medications that would prohibit participation in an exercise program

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Functional Assessment of Cancer Therapy Breast Symptom Index (FACT-B+4) Total Score from Baseline to 12 Weeks | Baseline and 12 weeks
  Assessed by the Functional Assessment of Cancer Therapy Breast Symptom Index (FACT-B+4), a 42-item measure of physical, emotional, social and functional well-being, as well as breast cancer specific symptomology associated with upper extremity dysfunction during the 7 days prior to questionnaire administration. Items are rated on a 5-point Likert-type scale with answers ranging from 0 "Not at all" to 4 "Very much." A total scores range is 0 to 168 with a higher score indicating better quality of life.

SECONDARY OUTCOMES:
Change in the Brief Pain Inventory Short Form (BPI SF) Score from Baseline to 12 Weeks | Baseline and 12 weeks
  Assessed by the Brief Pain Inventory Short Form (BPI SF), a 9-item measure of the severity of pain and pain interference in the 24 hour prior to questionnaire administrations. A simple numeric rating scale from 0 to 10 is used for item rating, and a total score is the mean of the item ratings. Higher scores indicate greater pain intensity and greater interference with function.
Change in the Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F) Total Score from Baseline to 12 Weeks | Baseline and 12 weeks
  Assessed by the Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F), a 13-item measure of the intensity of fatigue experienced during the 7 days prior to questionnaire administration. Items are rated on a 5-point Likert-type scale with answers ranging from 0 "Not at all" to 4 "very much" and items 7 and 8 being reversed score. A total scores range is 0 to 52 with a higher score indicating better quality of life.
Change in the Cancer Rehabilitation Evaluation Scale (CARES) Score from Baseline to 12 Weeks | Baseline and 12 weeks
  Assessed by the Cancer Rehabilitation Evaluation Scale (CARES), a 6-item measure of body image and self-esteem by measuring negative feelings about the body and self-perception in the month prior to questionnaire administration. Items are rated on a 5-point Likert-type scale with answers ranging from 0 "Not at all" to 4 "Very much." A total scores range is 0 to 24 with a higher score indicating greater negative body image and self-esteem.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu